CLINICAL TRIAL: NCT06491043
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study To Evaluate The Safety And Efficacy Of Umc119-06-05 Intravenous Infusion For The Treatment Of Subjects With Moderate To Severe Chronic Obstructive Pulmonary Disease
Brief Title: Treatment of Chronic Obstructive Pulmonary Disease by Infusion of Allogenic Mesenchymal Stem Cells
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Meribank Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UMC119-06-05-COPD-02
Record Dates: First submitted 2024-06-21; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized to one of the three groups: placebo control, low-dose allogeneic umbilical cord-derived mesenchymal stem cells UMC119-06-05 treatment, or high-dose UMC119-06-05 treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo (Placebo Comparator): normal saline, 4% human serum albumin
  Interventions: Other: UMC119-06-05
- low-dose UMC119-06-05 treatment (Experimental): normal saline, 4% human serum albumin, 1×10^8 cells/subject
  Interventions: Other: UMC119-06-05
- high-dose UMC119-06-05 treatment (Experimental): normal saline, 4% human serum albumin, 2×10^8 cells/subject
  Interventions: Other: UMC119-06-05

INTERVENTIONS:
Other: UMC119-06-05 — Human Umbilical Cord Derived-Mesenchymal Stem Cells

SUMMARY:
This phase II study is a randomized, placebo-controlled, double-blind study to evaluate the safety and efficacy of UMC119-06-05 compared to placebo in treating subjects with moderate to severe COPD. Eligible subjects will receive a single-dose IV infusion of UMC119-06-05 or placebo.

DETAILED DESCRIPTION:
Patients with chronic obstructive pulmonary disease (COPD) are characterized with airflow limitation and chronic inflammation, which is caused by cigarette smoking, noxious particles or gases. These inhaled irritants will induce inflammation, emphysema and fibrosis though chronic exposure. The current pharmacological treatment of COPD is symptomatic and is mainly based on bronchodilators and corticosteroids. Although current clinical treatment strategies can improve and stabilize COPD states and quality of life, none of them are able to modify the progressive decline in lung function, meaning it gradually gets worse over time. Therefore, development of new therapeutic modalities to improve the clinical outcomes and prognosis of COPD in adult patients is of urgent need. Among the more innovative, experimental therapies, mesenchymal stromal cells are proposed as a novel therapy with potential in treatment of COPD. This clinical trial is a phase II study. It is a randomized, placebo-controlled, double-blind study. Eligible subjects will be randomized to one of the three groups: placebo control, low-dose UMC119-06-05 treatment, or high-dose UMC119-06-05 treatment. Subjects will receive a single-dose IV infusion to evaluate the efficacy and long-term safety of UMC119-06-05 with moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Between ≥40 and ≤80 years of age, of either sex and of any race.
2. With diagnosis of COPD based on the Global Initiative for Chronic Obstructive Lung Disease (GOLD) standard.
3. Has a post-bronchodilator FEV1/FVC ratio <0.70.
4. Has a post-bronchodilator FEV1 predicted value ≥30% and <80%.
5. With a score ≥2 in the mMRC dyspnea scale.
6. With a score ≥10 in the COPD Assessment Test (CAT).
7. With a body weight ≥40 to ≤90 kg.
8. The disease status of COPD has been stable as determined by the investigator, and the standard treatment for COPD was not adjusted within 3 months prior to screening.
9. Is a current or ex-smoker, with a cigarette smoking history of ≥10 years or >10 pack-years.
10. Women of child-bearing potential should have a negative urine pregnancy test at screening, UNLESS they meet the following criteria:

(1)Post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with the serum follicle stimulating hormone (FSH) level >40 mIU/mL, OR; (2)6 weeks post-surgical bilateral oophorectomy with or without hysterectomy 11.Heterosexually active subjects must agree to use a double barrier method of birth control (or must have been surgically sterilized/post-menopausal) and not to donate sperms/eggs during the study.

12.Willing to provide written informed consent to participate in the study.

Exclusion Criteria:

1. Has evidence of active malignancy or prior history of active malignancy that has not been in complete remission for at least 5 years prior to screening.
2. Diagnosed with asthma or other clinically relevant lung disease other than COPD (e.g., restrictive lung diseases, sarcoidosis, tuberculosis, idiopathic pulmonary fibrosis, bronchiectasis, or lung cancer).
3. Has initiated pulmonary rehabilitation (e.g., exercise training) within 3 months prior to screening which, in the opinion of the Principal Investigator (PI), may affect the study's results.
4. Has documented history of uncontrolled heart failure.
5. Has pulmonary hypertension due to left heart condition.
6. Has atrial fibrillation or significant congenital heart defect/disease.
7. Has had a moderate or severe exacerbation of COPD (defined by GOLD standard) or has required mechanical ventilation (not including continuous positive airway pressure [CPAP]) within 30 days prior to screening.
8. Is hospitalized at screening.
9. With current active infection including pulmonary infection, systemic infection, or severe local infections.
10. Have the following conditions in laboratory tests at screening:

    1. >2 × upper limit of normal (ULN) for alanine aminotransferase (ALT) or aspartate aminotransferase (AST); or
    2. Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2; or
    3. White blood cells (WBC) <3.6 × 103/μL; or
    4. Platelet counts <150 × 103/μL; or
    5. Hemoglobin <10 g/dL; or
    6. Spot urine albumin-creatinine ratio (UACR) ≥30 mg/g; or
    7. Clinically significant hematuria or proteinuria deemed by the study investigator.
11. With known stage ≥3 chronic kidney disease.
12. Received systemic steroids or other immunosuppressants, immunomodulators, cytotoxic agents, chemotherapy, radiation therapy, or other cell therapies within 28 days or 5 half-lives, whichever is longer, prior to screening.
13. With known alpha-1 antitrypsin deficiency.
14. With known allergy or hypersensitivity to any component of the investigational product (IP) formulation (normal saline and human serum albumin [HSA]).
15. With a known history of drug-related anaphylaxis or other severe allergic reactions to drug.

    Note: "Severe" is defined as Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade 3 or greater.
16. Underwent major surgery (body organs that require anesthesia, such as tumor removal, open chest, heart surgery, abdominal surgery, intracranial surgery, or normal surgery for more than 3 hours, etc.) within 30 days prior to screening.
17. With known human immunodeficiency virus infection or immunocompromised.
18. With a known history of alcohol abuse or drug abuse within 5 years prior to screening.
19. Participating in another clinical study of new investigational therapies or have received an investigational therapy within 3 months prior to screening.
20. Pregnant (or plan to become pregnant within 3 months after study treatment) or lactating.
21. Has a life expectancy of <6 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From Baseline to Day 90]
  Incidence of any treatment-emergent serious adverse events (SAE), defined as the composite of: death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities.
  2.Incidence of related TEAEs and serious adverse events (SAEs) 3.Incidence of withdrawals due to adverse events (AEs) 4.Change/shift from baseline in laboratory tests 5.Change from baseline in vital signs 6.Shift from baseline in ECG results 7.Shift from baseline in physical examination results
Incidence of related TEAEs and serious adverse events (SAEs) | through the study
  Incidence of any treatment-emergent serious adverse events (SAE), defined as the composite of: death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities.
  2.Incidence of related TEAEs and serious adverse events (SAEs) 3.Incidence of withdrawals due to adverse events (AEs) 4.Change/shift from baseline in laboratory tests 5.Change from baseline in vital signs 6.Shift from baseline in ECG results 7.Shift from baseline in physical examination results
Incidence of withdrawals due to adverse events (AEs) | through the study
  AE incidence
Change/shift from baseline in laboratory tests | Baseline, 2 hours (h), Days 3, 7, 14, 28, 90
  laboratory tests
Change from baseline in vital signs | Baseline, 0 minute, 2 h, Days 3, 7, 14, 28, 90
  measure vital signs
shift from baseline in ECG results | Baseline, 2 h, Day 14
  ECG check
Shift from baseline in physical examination results | Baseline, 2 h, Days 3, 7, and 14
  physical examination

SECONDARY OUTCOMES:
Mean change from baseline in forced vital capacity (FVC) | Baseline, Days 28, 90, 180, 270, 360
  Respiratory functions (FVC) 2.Mean change from baseline in forced expiratory volume in one second (FEV1) 3.Mean change from baseline in FEV1/FVC ratio 4.Mean change from baseline in 6-minute walk test (6-MWT) 5.Mean change from baseline in St. George's Respiratory Questionnaire (SGRQ) score 6.Shift from baseline in modified Medical Research Council (mMRC) dyspnea scale 7.Incidence, frequency, and severity of COPD exacerbations 8.Time to first COPD exacerbation 9.Mean change or shift from baseline in Body mass index, airflow Obstruction, Dyspnea, and Exercise capacity (BODE) index 10.The number of times that rescue medication is used
Mean change from baseline in forced expiratory volume in one second (FEV1) | Baseline, Days 28, 90, 180, 270, 360
  Respiratory functions (FEV1)
Mean change from baseline in FEV1/FVC ratio | Baseline, Days 28, 90, 180, 270, 360
  Respiratory functions (FEV1/FVC)
Mean change from baseline in 6-minute walk test | Baseline, Days 28, 90, 180, 270, 360
  measure 6 minute walk distance
Mean change from baseline in St. George's Respiratory Questionnaire (SGRQ) score | Baseline, Days 28, 90, 180, 270, 360
  Georges Respiratory Questionnaire has scores range from 0 to 100, with higher scores indicating more limitations
Shift from baseline in modified Medical Research Council (mMRC) dyspnea scale | Baseline, Days 28, 90, 180, 270, 360
  mMRC dyspnea scale
Incidence, frequency, and severity of COPD exacerbations | through the study
  assess severity of COPD
Time to first COPD exacerbation | through the study
  assess severity and exacerbation
9. Mean change or shift from baseline in Body mass index, airflow Obstruction, Dyspnea, and Exercise capacity (BODE) index | baseline to Days 28, 90, 180, 270, 360
  BODE index
he number of times that rescue medication is used | through the study
  times of rescue medication

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, New Taipei City
  - Chang Gung Memorial Hospital, Linkou, Taoyuan

IPD SHARING:
Plan to Share IPD: No